CLINICAL TRIAL: NCT00709670
Title: ComParative Diagnostic Study Between MSCT and Stress Echography in Patients Presenting With Suspected Acute Coronary Syndrome Without ST Segment Elevation.
Brief Title: ComParative Diagnostic Study Between Multislice Computed Tomography (MSCT) and Stress Echography in Coronarin Patients.
Acronym: PEPSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P070607
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2008-07

CONDITIONS: Chest Pain
Keywords: MSCT; Echocardiography; Coronarography; Acute coronary syndrome without ST segment elevation; normal ECG; normal troponin; Acute
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- whole population who receive both tests (Experimental): this arm includes the whole study population who will receive both tests: MSCT and stress echocardiography
  Interventions: Procedure: MSCT and stress echocardiography

INTERVENTIONS:
Procedure: MSCT and stress echocardiography — tests MSCT and stress echocardiography
  Other Names: tests MSCT and stress echocardiography

SUMMARY:
The aim of this study is to define the best prognostic strategy for patients presenting suspected acute CORONARY syndrome, between MSCT and stress echocardiography.

DETAILED DESCRIPTION:
Patients presenting with a suspected acute CORONARY syndrome is based on the interrogation, the realization of an electrocardiogram (ECG) and 2 dosages of the cardiac troponin at some hours of interval. However, the ECG and the troponin are frequently normal and this does not absolutely eliminate the diagnosis. In that case, it is at present recommended to practise an effort ECG or a stress imaging, such as echocardiography. Several studies estimated the diagnostic exactness of stress echography for patients presenting a recent chest pain without modification of the ECG nor a rise of the troponin with a sensibility from 71 to 86% and a specificity from 91 to 98%. Recently, several teams estimated the interest of multislice computed tomography (MSCT) in the same population. The MSCT sensibility reported by 2 teams is promising because was found between 91 and 100%. On the other hand, the specificity was appreciably less good : between 76 and 82%. The negative predictive value to MSCT was excellent : between 97 and 100%.The aim of this work is to compare the diagnostic exactness between stress echography and MSCT for patients presenting with a suspected acute coronary syndrome without modification of the ECG nor rise of the troponin. It is about a prospective monocentric diagnostic study concerning 400 patients. The primary end point is the proportion report of true positives in MSCT with regard to stress echocardiography (the main diagnosis is the coronarography). The secondary end points include the proportion of false positives, the non interpretable or non contributory examination rate and especially the proportion of unwanted events in 6 months for the negative patients in both examinations according to a combined criteria including death, myocardial infraction (MI), percutaneous CORONARY intervention (PCI), coronary artery bypass graft (CABG) or readmission for chest pain with coronarography visualizing a stenosis greater than 50 %.

ELIGIBILITY:
Inclusion Criteria:

* chest pain < 24 hours
* normal ECG
* normal troponin I

Exclusion Criteria:

* ECG evolution
* troponin I evolution
* hemodynamic instability
* rhythmic instability
* allergy to iodized contrast products
* Creatinin > 150 micromol/L
* venous capital absence
* auricular fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Relative diagnostic accuracy of stress echography and MSCT at presentation of patients with acute chest pain and suspected acute coronary syndrome | 2 days

SECONDARY OUTCOMES:
proportion of AE in patients tested negative at both examinations: death, myocardial infraction, percutaneous coronary intervention, coronary artery bypass graft or readmission for chest pain with coronarography visualizing a stenosis greater than 50%. | 6 months
proportions of false positives, the reference method being coronarography. | 2 days
proportions of non interpretable or non contributory examinations | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric DURAND, MD PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hospital european Georges pompidou, Paris, France